CLINICAL TRIAL: NCT03135730
Title: International Rapid-onset Obesity with Hypothalamic Dysfunction, Hypoventilation, and Autonomic Dysregulation (ROHHAD) REDCap Registry
Brief Title: International Rapid-onset Obesity with Hypothalamic Dysfunction, Hypoventilation & Autonomic Dysregulation (ROHHAD) Registry
Status: Recruiting | Type: Observational
Sponsor: Debra Weese-Mayer (Other)
Collaborators: ROHHAD Fight Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Debra Weese-Mayer, Professor of Pediatric Autonomic Medicine, Northwestern University Feinberg School of Medicine Chief, Center for Autonomic Medicine in Pediatrics, Ann & Robert H. Lurie Children's Hospital of Chicago and Stanley Manne Children's Research Institute, Ann & Robert H Lurie Children's Hospital of Chicago
Organization: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Other Study IDs: 2012-14981 and 2013-15230b
Record Dates: First submitted 2017-04-27; First posted 2017-05-01 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-08

CONDITIONS: ROHHAD; Rapid-Onset Obesity with Hypothalamic Dysfunction, Hypoventilation & Autonomic Dysregulation
MeSH Terms: conditions — Hypoventilation; Primary Dysautonomias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: ROHHAD — Suspected and Confirmed ROHHAD cases

SUMMARY:
The Center for Autonomic Medicine in Pediatrics (CAMP) has collaborated with doctors from around the world to build the first International ROHHAD (Rapid-onset Obesity with Hypothalamic Dysfunction, Hypoventilation and Autonomic Dysregulation) REDCap (Research Electronic Data Capture) Registry. This registry is an international collaboration with ROHHAD patients and their physicians recruited from around the world.

The purpose of this IRB-approved research study is to gain a better understanding of the various health problems ROHHAD patients face with advancing age, and how these relate to each patient's specific medical course. With a better understanding of specific ROHHAD and associated clinical manifestations, we will be able to better anticipate healthcare needs and to provide more accurate guidelines to healthcare providers world-wide in caring for patients with ROHHAD.

The study aims to obtain detailed phenotypic information (information about health and well-being) on patients with ROHHAD. Participation would require filling out a confidential survey that asks questions regarding health and past medical history. Involvement in the project is completely voluntary and there is no compensation for taking part. However, this project will help us learn more about this devastating disease, with the goal of advancing treatment.

DETAILED DESCRIPTION:
ROHHAD is a rare, devastating disorder in which affected children demonstrate abnormalities of respiratory control, hypothalamic/endocrine function, and autonomic nervous system (ANS) dysregulation (ANSD). Affected children are seemingly normal until development of dramatic and rapid weight gain which occurs over a 6-month period between 1.5 and 10 years of age - heralding disease onset. The ROHHAD phenotype appears to evolve with advancing age and with variable timing of successive features. This study aims to develop a patient registry for ROHHAD, which will provide crucial insight into disease development, improving outcome in these children through improving early recognition of the disorder, understanding the phenotypic spectrum, and evolution of clinical course. Data will be stored in REDCap (Research Electronic Data Capture) system a secure web application designed exclusively to support data capture for research studies in a secure manner. The REDCap server is hosted securely at Northwestern University, behind a firewall, with virus protection, and using Secure Socket Layer (SSL) authentication to encrypt communication between a user and the server. Protected Health Information (PHI) will be labeled as such in the database and access to it will be restricted to the Principal Investigator (PI) and key personnel participating in the consent process and follow up contact of participants.

Participants in the International ROHHAD REDCap Registry will be identified and recruited from CAMP's registry of new, current, and past ROHHAD referrals, including ROHHAD patients referred for testing and/or consultation. Additionally, patients may also be recruited via the internet using emails, Facebook pages, and mailing lists for family groups. Anyone interested will be offered inclusion into the International ROHHAD Registry. Participants will be able to participate remotely, from their homes or locations where they have internet, phone, and computer access.

De-identified data collected through the REDCap registry will be de-identified and analyzed. Patients enrolled in this study will be offered participation in the NIH GRDR. This is an optional part of the study, and is not required for inclusion. The Global Rare Disease Registry (GRDR) is established by the NIH Office of Rare Disease Research. The goal of the GRDR is to establish a data repository of de-identified patient data, aggregated in a standardized manner, using Common Data Elements (CDEs) and standardized terminology. De-identification of patient's data will utilize the Global Unique Identifiers (GUID) system. Lurie Children's Hospital will retain ownership of all data shared with the GRDR. The de-identified data in the GRDR will be available to all investigators to enable analyses across many rare diseases and to facilitate various biomedical studies, including clinical trials, in pursuit of developing drugs and therapeutics to improve the healthcare and the quality of life for the many millions of people who are diagnosed with rare diseases.

Any patient agreeing to be part of the GRDR will have their data de-identified and this de-identified data exported and shared with the GRDR. These participants are also given the option to be contacted for participation in clinical trials. If this option is chosen, any researcher accessing de-identified information through the GRDR and planning to conduct a clinical trial will be allowed to contact the CAMP project coordinator to ask that patients fitting the profile of needed participants be contacted and offered inclusion. No de-identified information will be shared with researchers outside of CAMP, rather the CAMP project coordinator will contact identified patients fitting participation criteria to share contact information and details for the clinical trial. Interested patients will then be given to the option to contact researchers conducting clinical trials at their discretion.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of suspected ROHHAD
* Clinical diagnosis of confirmed ROHHAD

Exclusion Criteria:

* Clinical diagnosis not consistent with ROHHAD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected or confirmed ROHHAD worldwide
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-06-01 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2039-12-31 (Estimated)

PRIMARY OUTCOMES:
longitudinal clinical history in 200 ROHHAD patients | 10 years
  phenotype inclusive of control of breathing and autonomic regulation

SECONDARY OUTCOMES:
patient reported outcome measures to determine sensitive markers of disease progression or regression for use in intervention trials | 10 years
  phenotype inclusive of all systems served by the autonomic nervous system
patient registry for ROHHAD for use with the global rare diseases patient registry and data repository (GRDR) | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago and the Stanley Manne Children's Research Institute, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No